CLINICAL TRIAL: NCT00047177
Title: A Phase II Study of Oxaliplatin in Children With Recurrent or Refractory Medulloblastoma, Supratentorial Primitive Neuroectodermal Tumors and Atypical Teratoid Rhabdoid Tumors
Brief Title: Oxaliplatin in Treating Children With Recurrent or Refractory Medulloblastoma, Supratentorial Primitive Neuroectodermal Tumor, or Atypical Teratoid Rhabdoid Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James M. Boyett/PBTC Operations and Biostatistics Center Executive Director, Pediatric Brain Tumor Consortium
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000257562; PBTC-010
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent childhood medulloblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood ependymoma; childhood atypical teratoid/rhabdoid tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Medulloblastoma; Familial ependymoma; Rhabdoid Tumor | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of oxaliplatin in treating children who have recurrent or refractory medulloblastoma, supratentorial primitive neuroectodermal or atypical teratoid rhabdoid tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the objective response rate to oxaliplatin in pediatric patients with recurrent or refractory medulloblastoma at first progression.
* Estimate the objective response rate to oxaliplatin in pediatric patients with recurrent or refractory medulloblastoma at second or later relapse.
* Estimate the objective response rate to oxaliplatin in pediatric patients with recurrent or refractory supratentorial primitive neuroectodermal tumor, or atypical teratoid rhabdoid tumor.
* Describe the pharmacokinetics of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor type (medulloblastoma [measurable disease at first relapse vs positive cerebrospinal fluid or linear leptomeningeal disease vs measurable disease at second or later progression] vs supratentorial primitive neuroectodermal tumor vs atypical teratoid rhabdoid tumor).

Patients receive oxaliplatin IV over 2 hours on day 1. Treatment repeats every 21 days for up to 17 courses (1 year) in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 65 patients will be accrued for this study within 1.5-2.8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed medulloblastoma, supratentorial primitive neuroectodermal tumor (including pineoblastomas and ependymoblastomas), or atypical teratoid rhabdoid tumor

  * Recurrent or refractory disease
* Measurable disease by radiography
* Patients with positive cerebrospinal fluid cytology or linear leptomeningeal disease are eligible

PATIENT CHARACTERISTICS:

Age

* 21 and under

Performance status

* Karnofsky 50-100% OR
* Lansky 50-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3 (transfusion independent)
* Hemoglobin at least 8.0 g/dL (RBC transfusions allowed)

Hepatic

* Bilirubin no greater than 1.5 times normal
* ALT less than 2.5 times normal

Renal

* Creatinine no greater than 1.5 times normal OR
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min

Cardiovascular

* Shortening fraction at least 27% by echocardiogram OR
* Ejection fraction at least 50% by MUGA

Pulmonary

* No dyspnea at rest
* No exercise intolerance
* Pulse oximetry greater than 94%

Other

* No uncontrolled infection
* No active graft-versus-host disease
* No uncontrolled seizure disorders

  * Seizure disorders well controlled with anticonvulsants allowed
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 2 weeks since prior growth factors
* At least 6 months since prior allogeneic stem cell transplantation
* No concurrent colony-stimulating factors during the first course of study
* No concurrent immunomodulating agents

Chemotherapy

* At least 3 weeks since prior myelosuppressive therapy (6 weeks for nitrosoureas) and recovered
* No other concurrent anticancer chemotherapy

Endocrine therapy

* If concurrent corticosteroids necessary for intracranial pressure, must be on stable or decreasing dose for at least 1 week prior to study
* No other concurrent corticosteroids

Radiotherapy

* At least 2 weeks since prior local palliative radiotherapy (small port) to symptomatic metastatic sites
* At least 3 months since prior craniospinal radiotherapy
* No concurrent palliative radiotherapy
* Recovered from prior radiotherapy

Surgery

* Not specified

Other

* No other concurrent anticancer or experimental drugs

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2002-10; Primary Completion 2004-08 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Objective response rate to oxaliplatin in recurrent or progressive medulloblastoma at first progression
Objective response rate to oxaliplatin in recurrent or refractory medulloblastoma at second or later relapse

SECONDARY OUTCOMES:
Objective response rate to oxaliplatin in recurrent or progressive supratentorial PNETs or atypical teratoid rhabdoid tumor (ATRT)
Pharmacokinetics of oxaliplatin in the serum and CSF

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Fouladi, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (10):
- United States (10):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Fouladi M, Blaney SM, Poussaint TY, Freeman BB 3rd, McLendon R, Fuller C, Adesina AM, Hancock ML, Danks MK, Stewart C, Boyett JM, Gajjar A. Phase II study of oxaliplatin in children with recurrent or refractory medulloblastoma, supratentorial primitive neuroectodermal tumors, and atypical teratoid rhabdoid tumors: a pediatric brain tumor consortium study. Cancer. 2006 Nov 1;107(9):2291-7. doi: 10.1002/cncr.22241. PMID 17019740